CLINICAL TRIAL: NCT00421694
Title: Positive Surgical Margins Rate and EGFR Family Members Expression in Prostate Cancer Treated With Bicalutamide
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of L'Aquila (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SMBC142
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2007-10-08 (Estimated); Status verified 2007-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

INTERVENTIONS:
Drug: Bicalutamide

SUMMARY:
Following radical prostatectomy (RP), about 20% to 40% of the patients with prostate cancer (PCa) exhibit pathological parameters which are associated with a high risk of disease recurrence. The rationale for NHT is based on the theory that androgen ablation induces PCa apoptosis which induces a regression of the primary tumor bulk before RP. However the use of NHT prior RP is highly controversial. In spite of these unenthusiastic results, the relative short time of treatment and the use of different drugs from those utilized in other trials might still to make this regimen attractive in terms of drug related side effects and effectiveness. In this regard, Bicalutamide presents unique characteristics since it work differently respect to other anti-hormonal agents by interfering on both genotropic and non-genotropic mechanisms of androgen receptor

ELIGIBILITY:
Inclusion Criteria:

* Patients with cT2-T3a prostate cancer

Exclusion Criteria:

* Men>75 years
* Men<18 years
* Prior hormonal therapy
* Prior radiation or chemotherapy
* Prior investigational agents
* Life expectancy > 10 years
* Prior malignancy within the last five years
* Any other serious medical or psychiatric condition

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luca Gravina, M.D., Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Abruzzo, Italy